CLINICAL TRIAL: NCT00311246
Title: A Prospective Open-Label Trial of Adalimumab in Progressive Sarcoidosis
Brief Title: Trial of Adalimumab in Progressive Sarcoidosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruiting subjects
Sponsor: University of Chicago (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: University of Chicago #14093A
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-03

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Humira; Adalimumab; Tumor Necrosis Factor Inhibitors
MeSH Terms: conditions — Sarcoidosis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- An open-label (Experimental): Patients received adalimumab 40 mg weekly for 45 weeks, with a final follow-up at Week 52
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Subjects will give themselves a dose of Adalimumab at 40 mg/every week by subcutaneous injection for a total of 45 weeks.
  Other Names: Humira

SUMMARY:
Sarcoidosis is a rare disease that can affect any organ in the body. It is characterized by the buildup of immune-system (fights off infection in the body) cells in organs. These cells form small groups called granulomas, which lead to inflammation of the surrounding tissue. Sarcoidosis most commonly affects the lung and the lymph nodes (part of the immune system). The signs usually include shortness of breath, fever, dry cough, and chest pain. Other signs in many patients can include redness and painful lumps on the skin, reduced eyesight, joint pain, and rarely, nervous system damage. Sarcoidosis commonly affects young and middle-aged adults.

There are no approved therapies for the treatment of sarcoidosis. Corticosteroid (steroid hormone) therapy is considered the standard treatment. Only limited benefit has been shown when using corticosteroid therapy to ease lung symptoms or improve lung function in patients with sarcoidosis. Also, the effects of other therapies (for example: methotrexate, cyclophosphamide, anti-malarial drugs, thalidomide) and other immunosuppressants (drugs that suppress a body's natural defense system [immune system]) which have been used in a small number of patients are not well known and can cause long term problems.

The drug used in this study is called adalimumab. Adalimumab is FDA (Food and Drug Administration) approved for patients with moderately to severely active rheumatoid arthritis. However, adalimumab is not approved for the treatment of sarcoidosis. Adalimumab is experimental in this study. The purpose of this study is to evaluate the safety and effectiveness of adalimumab in the treatment of patients with sarcoidosis with pulmonary (lung) involvement who show symptoms of the disease even though they are currently being treated with medication.

DETAILED DESCRIPTION:
This study consists of 11 visits (including screening).

Screening Procedures:

A chest radiograph (PA and lateral) must be obtained within 3 months prior to the first study injection. It must indicate that subject is free of tuberculosis (TB). The chest radiograph will also be used to confirm the stage of the disease.

Histologically proven sarcoidosis will be confirmed.

Demographic data, a complete medical history (including signs and symptoms of sarcoidosis), a physical examination (including vital signs, weight and height). The medical history will include questions about history of recent TB and history of close contact with persons who might have TB. Concomitant medications, including the use of oral corticosteroids and immunosuppressants, will be reviewed and recorded. In addition the inclusion and exclusion criteria will be reviewed.

A tuberculin skin test will be performed.

A serum pregnancy test will be performed for all women within the 4-week period prior to the Baseline (Week 0) Visit. All women must test negative for pregnancy at screening.

ATS dyspnea score will be assessed.

The 6-minute walk test will be performed with Borg's CR10 dyspnea score obtained before and after.

Pulmonary function tests [PFTs] (spirometry) will be performed.

Blood samples for routine laboratory analyses will be obtained.

AE monitoring will also be performed.

Subjects who qualify for the study should be assigned to receive treatment within 14 days of the screening visit except if additional time is required for repeat TB skin testing.

Patients should still meet all of the inclusion criteria and none of the exclusion criteria at the time of the baseline visit before starting the injections. Subjects must agree to use appropriate contraception.

The procedures involved at all study visits are described below.

* Informed Consent:

(Screening Visit): Subjects will be asked to review this consent form and discuss with the study doctor or study staff any questions they may have

* Health and Medication Questions:

(Screen, Weeks 0, 2, 6, 12, 24, 30, 36, 45, 52): Subjects will be asked to answer questions about their health, their medical history, and the medications they take.

* Physical Exam:

(Screen, Weeks 6, 24, 52): Do a physical exam.

* Vital Signs:

(Screen, Weeks 0, 6, 12, 24, 52): Blood Pressure, Pulse, Temperature

* Height and Weight:

(Screen, Week 52)

* Blood Tests:

(Screen, Weeks 12, 24, 45, 52): Approximately 3 teaspoons of blood will be drawn from a vein in subject's hand or arm for these tests.

* Lung Function Test:

(Screen, Weeks 24, 52): Subject will be given a mouthpiece and asked to take deep breaths into a machine connected to a computer according to the cues of a staff member. The machine will measure the capacity of subject's lungs.

* Chest X-ray:

(Screen, Weeks 12, 24, 52):

* Tuberculosis Test:

(Screen only): Subject will be asked specific questions regarding their history of tuberculosis (also called TB: a type of bacterial lung infection) or personal contact with people with active tuberculosis. Subjects with active tuberculosis cannot be in the study. Subjects will be given a skin test for tuberculosis. For all subjects in this trial, a TB skin test with negative results must be obtained.

* 6 Minute Walk Test: (Screen, Weeks 0, 12, 24, 52): Subject will be asked to complete a test where they will walk for 6 minutes. Subject will be asked specific questions regarding any shortness of breath they have.
* Pregnancy Test:

(Screen only): A pregnancy blood test will be performed on all women of childbearing potential at the screening visit. The results of the test must be negative in order for subject to participate in the study.

* ECG:

(Week 0 only)

* Study Drug Administration:

(Weeks 0, 2, 6, 12, 18, 24, 30, 36, 45): Subject will receive study drug at the Week 0 Visit and be taught how to give themselves injections. Subject will be given a supply of study drug and clinical supplies that will last until the next study visit. Subject will be required to return all unused study drug as well as the packaging for the used study drug at each visit.

* Questionnaires:

(Weeks 0, 2, 12, 18, 24, 30, 36, 45): Prior to receiving any study drug, subject will be asked questions about their symptoms and quality of life, including their ability to care for themselves and carry out normal everyday activities (respiratory and health surveys) and health questionnaires.

All subjects will return for efficacy and safety evaluations at each time point including week 52, whether or not they complete the entire treatment schedule and whether or not they are (still) responding to treatment.

We will watch carefully for signs and symptoms of CHF and active TB at follow-up evaluations for all patients. The study agent will be stopped in subjects who are found to have NYHA Class III or IV CHF, severe right-sided heart failure, cor pulmonale, and/or active TB after enrollment in the study but they must return for further follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years of age.
* Sarcoidosis diagnosed at least 1 year prior to screening.
* Histologically proven sarcoidosis prior to screening.
* Have a diagnosis of sarcoidosis with evidence of parenchymal disease on chest radiograph (Stage II or III) or Stage I disease by chest radiographs and evidence of abnormal PFT as below or normal chest radiograph; or abnormal PFT, with abnormal chest computed tomography (CT) and evidence of sarcoid lung involvement by histology. Subjects with concurrent extrapulmonary sarcoidosis, particularly skin and eye involvement, are encouraged to be enrolled.
* Have forced vital capacity (FVC) > 40 and < 80% of predicted.
* Have an American Thoracic Society (ATS) dyspnea score of > Grade 1.
* Have been receiving pre-study treatment that includes at least 10 mg/day prednisone (or equivalent dose of corticosteroid) as a single agent, or 1 or more immunosuppressant (e.g., methotrexate, azathioprine, cyclophosphamide, chloroquine, leflunomide, hydroxychloroquine, mycophenolate mofetil, cyclosporine, tacrolimus, corticosteroids) for at least the 3-month period immediately prior to screening. Subjects must be on a stable dose of these medications for > 4 weeks before starting the study medication.
* Adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) must be used for the duration of the study and such precautions should be continued for 6 months after receiving the last study agent injection.
* Are considered eligible based on TB screening

Exclusion Criteria:

* Have used any investigational drug within 1 month prior to screening.
* Have received previous administration of a treatment with any other therapeutic agent targeted at reducing tumor necrosis factor [TNF] (e.g., pentoxifylline, thalidomide, etanercept, infliximab) within 3 months prior to screening.
* Have received previous administration of adalimumab.
* Have received any live virus or bacterial vaccinations within the 3 months before the first dose of the study agent or are expected to receive any live virus or bacterial vaccinations during the trial or up to 3 months after the last dose of the study agent.
* Have had any previous adverse reactions or allergic reactions (e.g., anaphylaxis) associated with the administration of monoclonal antibodies.
* Have New York Heart Association (NYHA) Class III or IV congestive heart failure (CHF).
* Have a history of severe right-sided heart failure or cor pulmonale.
* Have had serious infections within 2 months of screening. Less serious infections (such as acute upper respiratory tract infection [colds] or a simple urinary tract infection) need not be considered as exclusion at the discretion of the investigator.
* Are considered ineligible according to the United States of America (USA)-specific TB screening.
* Have or have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis and aspergilloma, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
* Have a known infection with human immunodeficiency virus (HIV).
* Have current signs and symptoms of systemic lupus erythematosus, or severe, progressive, or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic, or cerebral diseases (with the exception of sarcoidosis).
* Presence of a transplanted organ (with the exception of a corneal transplant) > 3 months prior to screening.
* Have any known malignancy or history of malignancy within 5 years prior to screening.
* Have a history of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease.
* Are pregnant, nursing, or planning pregnancy (both men and women) during the trial or within the 6-month period thereafter.
* Have had a known substance abuse or dependency, drug or alcohol within 3 years of screening.
* Have poor tolerability of subcutaneous injection or lack of adequate venous access for required blood sampling.
* Have a known history of demyelinating disease such as multiple sclerosis or optic neuritis.
* Presence of a non-sarcoidosis condition affecting survival.
* Have mental health problems interfering with participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-04; Primary Completion 2008-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadera J. Sweiss, M.D., Principal Investigator — The University of Chicago Hospitals
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Sweiss NJ, Noth I, Mirsaeidi M, Zhang W, Naureckas ET, Hogarth DK, Strek M, Caligiuri P, Machado RF, Niewold TB, Garcia JG, Pangan AL, Baughman RP. Efficacy Results of a 52-week Trial of Adalimumab in the Treatment of Refractory Sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 2014 Apr 18;31(1):46-54. PMID 24751453
- See also: Efficacy Results of a 52-week Trial of Adalimumab in the Treatment of Refractory Sarcoidosis. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4134103/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | An Open-label
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The population is male and female between the ages of 18-65
Arm/Group | An Open-label
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants] — YEARS IS A CATEGORICAL VARIABLE
  Participants
    <=18 years | 0
    Between 18 and 65 years | 11
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — THE UNIT OF MEASURE IS FEMALE, MALE
  Participants
    Female | 10
    Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in FVC From Screening to Week 24
Description: The forced vital capacity (FVC) measurement shows the amount of air a person can forcefully and quickly exhale after taking a deep breath. Improvement in FVC, if significant, means better breathing and lung function. The change in FVC done at screening and at week 24 were compared to notice if there were any changes.
Time Frame: 24 Weeks
Measure: Number; unit: Liters
Arm/Group | An Open-label
Number analyzed (Participants) | 11
Liters
  Participant 1 | -1
  Participant 2 | -3
  Participant 3 | 6
  Participant 4 | -1
  Participant 5 | -1
  Participant 6 | 4
  Participant 7 | 13
  Participant 8 | 5
  Participant 9 | 5
  Participant 10 | 3
  Participant 11 | -1

2. Secondary Outcome: Change in Distance Walked During 6 Minute Walk Test at Screening and 24 Weeks
Description: This is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes
Time Frame: 24 weeks
Measure: Number; unit: Meters
Arm/Group | An Open-label
Number analyzed (Participants) | 11
Meters
  Participant 1 | 124
  Participant 2 | -92
  Participant 3 | 20
  Participant 4 | 109
  Participant 5 | -34
  Participant 6 | 288
  Participant 7 | 124
  Participant 8 | -113
  Participant 9 | -44
  Participant 10 | 113
  Participant 11 | -90

3. Secondary Outcome: A Change in the Borg Dyspnea Score Before/After the 6 Minute Walk at Screening (S) and at 24 Weeks (W).
Description: This scale was used to measure a patients breathlessness before/after the 6 Minute Walk. This score was used at Screening (S) and at 24 weeks (W). The borg scale ranges from zero to 10 with zero being no breathlessness at all and 10 being maximal breathlessness. A change between screening and week 24 is reported.
Time Frame: 24 weeks
Measure: Number; unit: Units on a scale
Groups:
- Borg Dyspnea Scores: This scale was used to measure a patients breathlessness before/after the 6 Minute Walk at Screening and at 24 weeks.
Arm/Group | Borg Dyspnea Scores
Number analyzed (Participants) | 11
Units on a scale
  Participant 1 | 3
  Participant 2 | 3
  Participant 3 | 1
  Participant 4 | 3
  Participant 5 | 4
  Participant 6 | 0
  Participant 7 | 7.5
  Participant 8 | 2
  Participant 9 | 1.5
  Participant 10 | 0
  Participant 11 | 1

4. Secondary Outcome: Physicians Global Assessment of Disease Activity.
Description: This assessment to determine the level of disease activity. Scores range from 0 (no pulmonary manifestations of sarcoidosis) to 100 (worsening of pulmonary symptoms) on a visual analog scale.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physicians Global Assessment
Number analyzed (Participants) | 11
units on a scale | 81 (12)

5. Secondary Outcome: Patient's Global Assessment of Disease Activity.
Description: This is the patients measurement of disease activity. Scores range from 0 (no pulmonary manifestations of sarcoidosis) to 100 (worsening of pulmonary symptoms) on a visual analog scale.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients Global Assessment
Number analyzed (Participants) | 11
score on a scale | 54 (5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from week zero till week 52
Description: no serious adverse events
Groups:
- An Open-label: Patients received adalimumab 40 mg weekly for 45 weeks, with a final follow-up at Week 52
  Adalimumab: Subjects will give themselves a dose of Adalimumab at 40 mg/every week by subcutaneous injection for a total of 45 weeks.
  There were no adverse events.
Arm/Group | An Open-label
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No